CLINICAL TRIAL: NCT06731907
Title: KEYMAKER-U01 Substudy 01G: A Phase 2, Umbrella Study With Rolling Arms of Investigational Agents in Combination With Pembrolizumab With or Without Platinum-based Chemotherapy in Treatment-Naïve Participants With Stage IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Pembrolizumab With or Without Chemotherapy in Combination With Additional Treatments for Advanced Non-Small Cell Lung Cancer (NSCLC) (MK-3475-01G/KEYMAKER U01)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-01G; 2024-515772-12-00 (Registry Identifier: EU CT); U1111-1309-7532 (Registry Identifier: UTN); KEYMAKER U01 (Other: MSD); MK-3475-01G (Other: MSD)
Record Dates: First submitted 2024-12-11; First posted 2024-12-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Neoplasms; Lung Cancer; Pulmonary Neoplasms; Pulmonary Cancer; Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed; patritumab deruxtecan

STUDY DESIGN:
Intervention Model Description: This is a multi site, rolling-arm study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab and Chemotherapy (Active Comparator): Pembrolizumab will be administered as a 200mg IV infusion on Day 1 of every three weeks (Q3W) for up to 35 cycles (~ 2 years). The doublet platinum-based chemotherapy treatments used in this substudy are standard-of care regimens for squamous (paclitaxel/Nab-paclitaxel and carboplatin) and nonsquamous (pemetrexed and carboplatin) NSCLC. Pemetrexed is administered as a 500mg/m^2 IV infusion Q3W until discontinuation criterion is met. Nab-paclitaxel will be administered as a 100mg/m^2 IV infusion on Days 1, 8, and 15 Q3W for up to 4 cycles. Paclitaxel will be administered as a 200 mg/m^2 IV infusion on Day 1 Q3W for up to 4 cycles. Carboplatin will be administered as an IV infusion area under the time x concentration curve (AUC) for 4 cycles as per local practice and labels. The dose will be AUC5 or 6 mg/mL•min Q3W and will not exceed 900mg.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Pemetrexed
- Pembrolizumab and HER3-DXd (Experimental): Pembrolizumab will be administered as a 200mg IV infusion on Day 1 Q3W for up to 35 cycles (~ 2 years). HER3-Dxd will be administered as 5.6mg/kg IV infusion on Day 1 Q3W until discontinuation criteria is met.
  Interventions: Biological: Pembrolizumab; Biological: HER3-DXd

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 200mg IV Infusion.
  Other Names: Keytruda®, MK-3475, SCH 900475
Drug: Carboplatin — Carboplatin IV infusion AUC5 or 6 mg/mL•min and not exceeding 900mg.
  Other Names: Paraplatin®
  Arms: Pembrolizumab and Chemotherapy
Drug: Paclitaxel — Paclitaxel 200 mg/m^2 IV infusion.
  Other Names: Taxol
  Arms: Pembrolizumab and Chemotherapy
Drug: Nab-paclitaxel — Nab-paclitaxel 100mg/m^2 IV infusion.
  Other Names: Abraxane
  Arms: Pembrolizumab and Chemotherapy
Drug: Pemetrexed — Pemetrexed 500mg/m^2 IV infusion.
  Other Names: Alimta
  Arms: Pembrolizumab and Chemotherapy
Biological: HER3-DXd — HER3-Dxd 5.6mg/kg IV infusion.
  Other Names: patritumab deruxtecan, U3-1402, MK-1022
  Arms: Pembrolizumab and HER3-DXd

SUMMARY:
Researchers are investigating new treatments for untreated advanced non-small cell lung cancer (NSCLC), which is the most common form of lung cancer and lung cancer that has spread beyond surgical removal. Standard treatments include immunotherapy, such as pembrolizumab, and chemotherapy. This study aims to determine the effectiveness of adding other treatments, including the human epidermal growth factor receptor 3-directed antibody-drug conjugate (HER3-DXd) patritumab deruxtecan, to pembrolizumab, with or without chemotherapy. The primary goals are to assess safety and efficacy of the treatments.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Histologically or cytologically confirmed diagnosis of Stage IV squamous or non-squamous non-small cell lung cancer (NSCLC) per American Joint Committee on Cancer (AJCC) Staging Manual Version 8.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1 as assessed within 7 days before randomization.
* Has archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated has been provided.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on ART.
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to treatment randomization.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements.
* Participants with squamous histology are excluded if there is a known tumor-activating epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) or c ros oncogene 1 (ROS1) gene rearrangement.
* Is HIV-infected with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, or any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement.
* Has evidence of any leptomeningeal disease.
* Has known history of, or active, neurologic paraneoplastic syndrome.
* Has clinically significant corneal disease.
* Has myocardial infarction within 6 months.
* Has New York Heart Association (NYHA) Classes 3 or 4 congestive heart failure.
* Has uncontrolled angina pectoris within 6 months.
* Has cardiac arrhythmia requiring ongoing antiarrhythmic treatment.
* Has history of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes.
* Has bradycardia of less than 50 beats per minute (bpm) unless the participant has a pacemaker.
* Has history of second- or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers and have no history of fainting or clinically relevant arrhythmia with pacemakers.
* Has coronary/peripheral artery bypass graft within 6 months.
* Has complete left bundle branch block.
* Has inadequate washout period from prior concomitant therapy as specified in protocol before randomization.
* Has received prior treatment with a topoisomerase I inhibitor or an anti-HER3 antibody and/or ADC that consists of an exatecan derivative that is a topoisomerase I inhibitor.
* Has received prior systemic anticancer therapy for their metastatic NSCLC.
* Has received prior therapy with an anti- programmed cell death 1 protein (anti-PD-1), anti- programmed cell death ligand 1 protein (anti-PD-L1), or anti- programmed cell death ligand 2 protein (anti-PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor.
* Has received prior radiotherapy within 2 weeks of randomization, has radiation related toxicity requiring corticosteroids, or has had radiation pneumonitis.
* Has received radiation therapy to the lung that is >30 gray within 6 months of start of study intervention.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity to any of the study interventions and/or any of their excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has active infection requiring systemic therapy.
* Has concurrent active Hepatitis B and Hepatitis C virus infection.
* Have not adequately recovered from major surgery or have ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2032-03-12 (Estimated); Study Completion 2032-03-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to ~ 5 years
  ORR is defined as a confirmed complete response or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by Blinded Independent Central Review (BICR).
Number of Participants with Adverse Events (AEs) | Up to ~ 5 years
  Adverse events are any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Number of Participants Discontinuing Study Drug Due to AEs | Up to ~ 2 years
  Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to ~ 5 years
  For participants who demonstrate a confirmed complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by BICR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) | Up to ~ 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by BICR or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to ~ 5 years
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (40):
- United States (5):
  - University of Kentucky ( Site 0019), Lexington, Kentucky
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
  - Sanford Fargo Medical Center ( Site 0039), Fargo, North Dakota
  - Abramson Cancer Center ( Site 0010), Philadelphia, Pennsylvania
  - Sanford Cancer Center ( Site 0038), Sioux Falls, South Dakota
- Chile (3):
  - Centro de Estudios Clínicos SAGA ( Site 0162), Santiago, Region M. de Santiago
  - FALP ( Site 0161), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0160), Santiago, Region M. de Santiago
- Greece (2):
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 0204), Athens, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 0205), Thessaloniki
- Hungary (3):
  - Petz Aladar Egyetemi Oktato Korhaz ( Site 0062), Győr, Győr-Moson-Sopron
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Gyula Korhaz-Rendelointezet ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
  - Országos Korányi Pulmonológiai Intézet ( Site 0060), Budapest
- Israel (6):
  - Rambam Health Care Campus ( Site 0076), Haifa
  - Shaare Zedek Medical Center ( Site 0075), Jerusalem
  - Meir Medical Center ( Site 0071), Kfar Saba
  - Rabin Medical Center ( Site 0074), Petah Tikva
  - Sheba Medical Center ( Site 0070), Ramat Gan
  - Sourasky Medical Center ( Site 0077), Tel Aviv
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0175), Milan, Lombardy
  - IRCCS Ospedale San Raffaele ( Site 0171), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 0174), Roma
- Poland (4):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii-Oddzial Onkologii Klinicznej z Pododdzialem Dz ( Site 0153), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0152), Koszalin, West Pomeranian Voivodeship
- Spain (3):
  - Institut Català d'Oncologia - L'Hospitalet ( Site 0090), L'Hospitalet de Llobregat, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 0092), Barcelona
  - Hospital Universitario Quiron Madrid ( Site 0091), Madrid
- Taiwan (2):
  - Taipei Medical University Hospital ( Site 0180), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0182), Taoyuan District
- Turkey (Türkiye) (3):
  - Baskent University Dr. Turgut Noyan Research and Training Center ( Site 0141), Adana
  - Hacettepe Universite Hastaneleri ( Site 0140), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 0142), Ankara
- Ukraine (6):
  - CNE CC of Oncology Hematol ( Site 0130), Cherkasy, Cherkasy Oblast
  - Municipal Enterprise "Bukovinian сlinical oncology сenter" ( Site 0136), Chernivtsi, Chernivetska Oblast
  - CNCE Precarpathian Clinical Oncologic Center ( Site 0131), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - VISION PARTNER Medical Centre ( Site 0134), Kyiv, Kyivska Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council" ( Site 0133), Vinnytsia, Vinnytsia Oblast
  - Shalimov Institute of Surgery and Transplantation ( Site 0135), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26442&tenant=MT_MSD_9011